CLINICAL TRIAL: NCT01238211
Title: A Phase II Study of Induction (Daunorubicin/Cytarabine) and Consolidation (High-Dose Cytarabine) Chemotherapy Plus Dasatinib (NSC #732517) and Continuation Therapy With Dasatinib Alone in Newly Diagnosed Patients With Core Binding Factor Acute Myeloid Leukemia (AML)
Brief Title: Combination Chemotherapy and Dasatinib in Treating Patients With Newly Diagnosed Acute Myeloid Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-02615; NCI-2011-02615 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000688434; CALGB-10801 (Other: Alliance for Clinical Trials in Oncology); CALGB-10801 (Other: CTEP); U10CA180821 (NIH); U10CA031946 (NIH)
Record Dates: First submitted 2010-11-09; First posted 2010-11-10 (Estimated); Results first posted 2014-08-12 (Estimated); Last update posted 2023-03-01 (Actual); Status verified 2023-01

CONDITIONS: Acute Myeloid Leukemia; Acute Myeloid Leukemia Arising From Previous Myelodysplastic Syndrome; Adult Acute Myeloid Leukemia With Inv(16)(p13.1q22); CBFB-MYH11; Adult Acute Myeloid Leukemia With t(16;16)(p13.1;q22); CBFB-MYH11; Adult Acute Myeloid Leukemia With t(8;21); (q22; q22.1); RUNX1-RUNX1T1; Core Binding Factor Acute Myeloid Leukemia; Secondary Acute Myeloid Leukemia; Therapy-Related Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia, Myelomonocytic, Acute | interventions — Cytarabine; Dasatinib; Daunorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (daunorubicin hydrochloride, cytarabine, dasatinib) (Experimental): INDUCTION THERAPY (course 1): Patients receive daunorubicin hydrochloride IV on days 1-3, cytarabine IV continuously over 168 hours on days 1-7, and dasatinib PO QD on days 8-21. Patients with responsive disease on day 21 undergo consolidation therapy, and patients with non-responsive disease on day 21 (bone marrow cellularity >= 20% and leukemia blasts >= 5%) receive a second course of induction therapy.
  INDUCTION THERAPY (course 2): Patients receive daunorubicin hydrochloride IV on days 1-3, cytarabine IV continuously over 120 hours on days 1-5, and dasatinib PO QD on days 6-19. Patients achieving complete response receive consolidation therapy.
  CONSOLIDATION THERAPY: Patients receive high-dose cytarabine IV over 3 hours on days 1, 3, and 5, and dasatinib PO QD on days 6-26 or 7-27. Treatment repeats every 28 days for up to 4 courses in the absence of disease progression or unacceptable toxicity. Patients in complete remission receive continuation therapy.
  Interventions: Drug: Cytarabine; Drug: Dasatinib; Drug: Daunorubicin Hydrochloride; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Cytarabine — Given IV
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-Cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Drug: Dasatinib — Given PO
  Other Names: BMS-354825; Dasatinib Hydrate; Dasatinib Monohydrate; Sprycel
Drug: Daunorubicin Hydrochloride — Given IV
  Other Names: Cerubidin; Cerubidine; Cloridrato de Daunorubicina; Daunoblastin; Daunoblastina; Daunoblastine; Daunomycin Hydrochloride; Daunomycin, hydrochloride; Daunorubicin.HCl; Daunorubicini Hydrochloridum; FI-6339; Ondena; RP-13057; Rubidomycin Hydrochloride; Rubilem
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase II trial studies the side effects and how well giving combination chemotherapy together with dasatinib works in treating patients with newly diagnosed acute myeloid leukemia. Drugs used in chemotherapy, such as daunorubicin hydrochloride and cytarabine, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Dasatinib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Giving combination chemotherapy together with dasatinib may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the safety and tolerability of dasatinib 100 mg/day given after intensive induction (daunorubicin hydrochloride [daunorubicin]/cytarabine), and consolidation chemotherapy (high-dose cytarabine) and as single agent in maintenance therapy to newly diagnosed patients with core binding factor acute myeloid leukemia (AML).

II. 30-day survival rate during induction (the lack of early/hypoplastic death).

III. The absence of pleural or pericardial effusion, and absence of liver toxicity that exceeds grade 2.

SECONDARY OBJECTIVES:

I. To assess clinical outcomes such as event-free survival (EFS), complete response (CR) rate, cumulative incidence of relapse (CIR), cumulative incidence of death (CID), disease-free survival (DFS), and overall survival (OS).

II. To describe the frequency and severity of adverse events of patients treated on this study during induction, consolidation, and continuation therapy.

III. To describe the interaction of pretreatment disease and patient characteristics including morphology, cytogenetics, immunophenotype, molecular genetic features, white blood cell (WBC) count and hemogram, and performance status on clinical outcomes.

OUTLINE:

INDUCTION THERAPY (course 1): Patients receive daunorubicin hydrochloride intravenously (IV) on days 1-3, cytarabine IV continuously over 168 hours on days 1-7, and dasatinib orally (PO) once daily (QD) on days 8-21. Patients with responsive disease on day 21 undergo consolidation therapy, and patients with non-responsive disease on day 21 (bone marrow cellularity >= 20 % and leukemia blasts >= 5%) receive a second course of induction therapy.

INDUCTION THERAPY (course 2): Patients receive daunorubicin hydrochloride IV on days 1-3, cytarabine IV continuously over 120 hours on days 1-5, and dasatinib PO once a day on days 6-19. Patients achieving complete response receive consolidation therapy.

CONSOLIDATION THERAPY: Patients receive high-dose cytarabine IV over 3 hours on days 1, 3, and 5, and dasatinib PO QD on days 6-26 or 7-27. Treatment repeats every 28 days for up to 4 courses in the absence of disease progression or unacceptable toxicity. Patients in complete remission receive continuation therapy.

CONTINUATION THERAPY: Patients receive dasatinib PO on days 1-28. Treatment repeats every 28 days for 12 courses in the absence of disease progression or unacceptable toxicity.

After completion of study therapy, patients are followed up every 2 months for 2 years, every 3 months for 2 years, and then every year for up to 10 years from study entry.

ELIGIBILITY:
Inclusion Criteria:

* Documentation of disease as assessed by the Alliance reference laboratory at the Ohio State University per Cancer and Leukemia Group B (CALGB) 20202, molecular diagnosis of core-binding factor (CBF) acute myeloid leukemia (AML) by reverse transcriptase polymerase chain reaction (RT-PCR) positive for RUNX1-RUNX1T1 fusion transcript resulting from t(8;21)(q22;q22) (or a variant form) or CBFB-MYH11 fusion transcript resulting from inv(16)(p13.1q22) or t(16;16)(p13.1;q22) (any % bone marrow or blood blasts render the diagnosis of CBF AML based on the World Health Organization [WHO] classification)
* No prior chemotherapy for leukemia or myelodysplasia with the following exceptions:

  * Emergency leukapheresis
  * Emergency treatment for hyperleukocytosis with hydroxyurea,
  * Cranial radiotherapy (RT) for central nervous system (CNS) leukostasis (one dose only),
  * Growth factor/cytokine support/non-cytotoxic molecular-targeted agents
* AML patients with a history of antecedent myelodysplasia (MDS) remain eligible for treatment on this trial
* Patients who have developed therapy related myeloid neoplasm (t-MN) after prior radiation therapy or chemotherapy for another cancer or disorder are eligible
* Left ventricular ejection fraction >= lower limit of institutional normal by multigated acquisition (MUGA) or echocardiogram (ECHO) scan
* Patients must not have had myocardial infarction within 6 months of registration
* Patients must not have had ventricular tachyarrhythmia within 6 months of registration
* Patients must have no major conduction abnormality (unless a cardiac pacemaker is present)
* Bilirubin must not be < 2.5 times upper limit of normal
* Patients must be non-pregnant and non-nursing; pregnant or nursing patients may not be enrolled; women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test within a sensitivity of at least 25 mIU/mL within 72 hours prior to registration; women of child-bearing potential must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control - one highly effective method (e.g., intrauterine device [IUD], hormonal, tubal ligation, or partner's vasectomy), and one additional effective method (e.g., latex condom, diaphragm, or cervical cap) - AT THE SAME TIME, before she begins dasatinib therapy, during treatment and at least 12 weeks after treatment is complete; "Women of childbearing potential" is defined as a sexually active mature woman who has not undergone a hysterectomy or who has had menses at any time in the preceding 24 consecutive months
* Patients with congenital long QT syndrome or non-congenital corrected QT (QTc) prolongation (defined as a QTc interval consistently equal to or greater than 480 msecs) that cannot be corrected by infusion of electrolytes and/or discontinuation of other medications prior to start of treatment are excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2010-12-14 (Actual); Primary Completion 2013-07-01 (Actual); Study Completion 2021-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guido Marcucci, Principal Investigator — Alliance for Clinical Trials in Oncology
Locations (65):
- United States (65):
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - AdventHealth Orlando, Orlando, Florida
  - Saint Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Graham Hospital Association, Canton, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital, Carthage, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Heartland Cancer Research NCORP, Decatur, Illinois
  - Eureka Hospital, Eureka, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Mason District Hospital, Havana, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Mcdonough District Hospital, Macomb, Illinois
  - Bromenn Regional Medical Center, Normal, Illinois
  - Carle Cancer Institute Normal, Normal, Illinois
  - Illinois CancerCare-Community Cancer Center, Normal, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Ottawa Regional Hospital and Healthcare Center, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin Cancer Treatment Center, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois Valley Hospital, Peru, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - Illinois CancerCare-Spring Valley, Spring Valley, Illinois
  - Fort Wayne Medical Oncology and Hematology Inc-Parkview, Fort Wayne, Indiana
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - Eastern Maine Medical Center, Bangor, Maine
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Christiana Care - Union Hospital, Elkton, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Bronson Battle Creek, Battle Creek, Michigan
  - Spectrum Health Big Rapids Hospital, Big Rapids, Michigan
  - Cancer Research Consortium of West Michigan NCORP, Grand Rapids, Michigan
  - Mercy Health Saint Mary's, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Mercy Health Mercy Campus, Muskegon, Michigan
  - Spectrum Health Reed City Hospital, Reed City, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - University of Missouri - Ellis Fischel, Columbia, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Northwell Health NCORP, Lake Success, New York
  - Northwell Health/Center for Advanced Medicine, Lake Success, New York
  - North Shore University Hospital, Manhasset, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Central Vermont Medical Center/National Life Cancer Treatment, Berlin Corners, Vermont
  - University of Vermont and State Agricultural College, Burlington, Vermont

REFERENCES:
- [Derived] Marcucci G, Geyer S, Laumann K, Zhao W, Bucci D, Uy GL, Blum W, Eisfeld AK, Pardee TS, Wang ES, Stock W, Kolitz JE, Kohlschmidt J, Mrozek K, Bloomfield CD, Stone RM, Larson RA. Combination of dasatinib with chemotherapy in previously untreated core binding factor acute myeloid leukemia: CALGB 10801. Blood Adv. 2020 Feb 25;4(4):696-705. doi: 10.1182/bloodadvances.2019000492. PMID 32092139
- [Derived] Yin J, LaPlant B, Uy GL, Marcucci G, Blum W, Larson RA, Stone RM, Mandrekar SJ. Evaluation of event-free survival as a robust end point in untreated acute myeloid leukemia (Alliance A151614). Blood Adv. 2019 Jun 11;3(11):1714-1721. doi: 10.1182/bloodadvances.2018026112. PMID 31171508

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between April 2011 and January 2013, 61 participants were recruited.
Groups:
- Treatment (Daunorubicin Hydrochloride, Cytarabine, Dasatinib): INDUCTION THERAPY: daunorubicin hydrochloride IV (60 mg/m^2)on days 1-3, cytarabine IV (200 mg/m^2) continuously over 168 hours on days 1-7, and dasatinib PO (100 mg) once daily on days 8-21. Patients achieving a response go to consolidation therapy, and patients not achieving a receive a second course of induction therapy.
  CONSOLIDATION THERAPY: high-dose cytarabine IV (patients < Age 60: 3000 mg/m^2, Age >= 1000 mg/m^2)over 3 hours on days 1, 3, and 5, and dasatinib PO (100 mg) once daily on days 6-26. Treatment repeats every 28 days for 4 courses in the absence of disease progression or unacceptable toxicity. Patients in complete remission receive continuation therapy.
  CONTINUATION THERAPY: dasatinib PO (100 mg) once daily for 12 months or relapse.
Period: Overall Study
Arm/Group | Treatment (Daunorubicin Hydrochloride, Cytarabine, Dasatinib)
Started | 61
Completed | 3
Not Completed | 58
Not completed — Continues active treatment | 31
Not completed — Adverse Event | 7
Not completed — Death | 4
Not completed — Relapse/Progression | 2
Not completed — Withdrawal by Subject | 7
Not completed — Non-protocol treatment | 4
Not completed — Investigator/Patient Decision | 3

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Daunorubicin Hydrochloride, Cytarabine, Dasatinib)
Number analyzed (Participants) | 61
Age, Continuous [Median (Full Range); unit: years] | 51 [19.8 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 54
  Unknown or Not Reported | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 5
  White | 46
  More than one race | 0
  Unknown or Not Reported | 8
Region of Enrollment [Number; unit: participants]
  United States | 61

OUTCOME MEASURES:

1. Primary Outcome: 30 Day Survival Rate
Description: Percentage of participants who were alive 30 days after starting induction treatment.
Time Frame: 30 days
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Daunorubicin Hydrochloride, Cytarabine, Dasatinib)
Number analyzed (Participants) | 61
percentage of participants | 97 [89 to 99.6]

2. Secondary Outcome: Event-free Survival
Description: Event free survival (EFS) is defined as the time from registration to failure to achieve complete remission (CR), relapse after CR is attained or death, whichever comes first. The 1 year EFS rate with 95% CI was estimated using the Kaplan-Meier method,
  Complete remission (CR) is defined as: disappearance of all clinical and/or radiologic evidence of disease. Neutrophil count > 1.0 x 10^9/L and platelet count > 100 x 10^9/L, and normal bone marrow differential (< 5% blasts).
Time Frame: 1 year
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Treatment (Daunorubicin Hydrochloride, Cytarabine, Dasatinib)
Number analyzed (Participants) | 61
percentage of patients | 83 [70.7 to 90.5]

3. Secondary Outcome: Complete Response Rate
Description: Percentage of participants who achieve a CR. Complete remission (CR) is defined as: disappearance of all clinical and/or radiologic evidence of disease. Neutrophil count > 1.0 x 10^9/L and platelet count > 100 x 10^9/L, and normal bone marrow differential (< 5% blasts).
Time Frame: 60 months
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Treatment (Daunorubicin Hydrochloride, Cytarabine, Dasatinib)
Number analyzed (Participants) | 61
percentage of patients | 90 [80 to 96]

4. Secondary Outcome: Cumulative Incidence of Relapse
Time Frame: 60 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Daunorubicin Hydrochloride, Cytarabine, Dasatinib)
Number analyzed (Participants) | 61
Participants | 10

5. Secondary Outcome: Cumulative Incidence of Death
Time Frame: 36 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Daunorubicin Hydrochloride, Cytarabine, Dasatinib)
Number analyzed (Participants) | 61
Participants | 15

6. Secondary Outcome: Disease-free Survival
Description: Disease free survival (DFS) is defined as the time from achievement of CR to relapse or death, whichever comes first. The 3 year DFS rate with 95% CI was estimated using the Kaplan-Meier method.
Time Frame: 3 years
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Treatment (Daunorubicin Hydrochloride, Cytarabine, Dasatinib)
Number analyzed (Participants) | 61
percentage of patients | 75 [63 to 89]

7. Secondary Outcome: Overall Survival
Description: Overall survival (OS) is defined as time from registration to death. The 3 year OS rate with 95% CI was estimated using the Kaplan-Meier method.
Time Frame: 3 years
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Treatment (Daunorubicin Hydrochloride, Cytarabine, Dasatinib)
Number analyzed (Participants) | 61
percentage of patients | 77 [66 to 89]

ADVERSE EVENTS:
Time Frame: 3 years
Groups:
- Treatment (Daunorubicin Hydrochloride, Cytarabine, Dasatinib): CONTINUATION THERAPY: dasatinib PO (100 mg) once daily for 12 months or relapse.
Arm/Group | Treatment (Daunorubicin Hydrochloride, Cytarabine, Dasatinib)
All-Cause Mortality (participants affected / at risk) | 15/61
Serious Adverse Events (participants affected / at risk) | 27/61
Other Adverse Events (participants affected / at risk) | 61/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Daunorubicin Hydrochloride, Cytarabine, Dasatinib) (N=61)
Anemia (Blood and lymphatic system disorders) | 26
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 2
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 18
Atrial fibrillation (Cardiac disorders) | 2
Atrial flutter (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 1
Chest pain - cardiac (Cardiac disorders) | 2
Palpitations (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 11
Supraventricular tachycardia (Cardiac disorders) | 1
Ventricular arrhythmia (Cardiac disorders) | 1
Ventricular tachycardia (Cardiac disorders) | 2
Hyperthyroidism (Endocrine disorders) | 1
Blurred vision (Eye disorders) | 1
Conjunctivitis (Eye disorders) | 1
Dry eye (Eye disorders) | 1
Eye disorders - Other (Eye disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 4
Ascites (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 6
Dental caries (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 13
Dyspepsia (Gastrointestinal disorders) | 2
Dysphagia (Gastrointestinal disorders) | 1
Fecal incontinence (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 3
Gastrointestinal pain (Gastrointestinal disorders) | 1
Hemorrhoids (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 20
Oral hemorrhage (Gastrointestinal disorders) | 1
Oral pain (Gastrointestinal disorders) | 2
Toothache (Gastrointestinal disorders) | 1
Typhlitis (Gastrointestinal disorders) | 1
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 13
Chills (General disorders) | 5
Edema face (General disorders) | 1
Edema limbs (General disorders) | 5
Edema trunk (General disorders) | 2
Fatigue (General disorders) | 22
Fever (General disorders) | 9
General disorders and administration site conditions - Other (General disorders) | 5
Infusion related reaction (General disorders) | 1
Malaise (General disorders) | 3
Multi-organ failure (General disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Pain (General disorders) | 5
Hepatic hemorrhage (Hepatobiliary disorders) | 1
Catheter related infection (Infections and infestations) | 2
Enterocolitis infectious (Infections and infestations) | 1
Infections and infestations - Other (Infections and infestations) | 3
Lung infection (Infections and infestations) | 8
Mucosal infection (Infections and infestations) | 2
Sepsis (Infections and infestations) | 6
Sinusitis (Infections and infestations) | 1
Skin infection (Infections and infestations) | 2
Small intestine infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Bruising (Injury, poisoning and procedural complications) | 2
Fall (Injury, poisoning and procedural complications) | 1
Activated partial thromboplastin time prolonged (Investigations) | 9
Alanine aminotransferase increased (Investigations) | 15
Alkaline phosphatase increased (Investigations) | 9
Aspartate aminotransferase increased (Investigations) | 17
Blood bilirubin increased (Investigations) | 10
Cardiac troponin I increased (Investigations) | 1
Creatinine increased (Investigations) | 11
Electrocardiogram QT corrected interval prolonged (Investigations) | 6
Hemoglobin increased (Investigations) | 1
INR increased (Investigations) | 9
Investigations - Other (Investigations) | 3
Lymphocyte count decreased (Investigations) | 18
Lymphocyte count increased (Investigations) | 2
Neutrophil count decreased (Investigations) | 26
Platelet count decreased (Investigations) | 27
Weight gain (Investigations) | 1
Weight loss (Investigations) | 6
White blood cell decreased (Investigations) | 18
Acidosis (Metabolism and nutrition disorders) | 4
Alkalosis (Metabolism and nutrition disorders) | 2
Anorexia (Metabolism and nutrition disorders) | 11
Dehydration (Metabolism and nutrition disorders) | 3
Hyperglycemia (Metabolism and nutrition disorders) | 19
Hyperkalemia (Metabolism and nutrition disorders) | 7
Hypermagnesemia (Metabolism and nutrition disorders) | 3
Hypernatremia (Metabolism and nutrition disorders) | 4
Hyperuricemia (Metabolism and nutrition disorders) | 6
Hypoalbuminemia (Metabolism and nutrition disorders) | 21
Hypocalcemia (Metabolism and nutrition disorders) | 12
Hypoglycemia (Metabolism and nutrition disorders) | 3
Hypokalemia (Metabolism and nutrition disorders) | 16
Hypomagnesemia (Metabolism and nutrition disorders) | 6
Hyponatremia (Metabolism and nutrition disorders) | 13
Hypophosphatemia (Metabolism and nutrition disorders) | 6
Metabolism and nutrition disorders - Other (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 4
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Ataxia (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 5
Dysgeusia (Nervous system disorders) | 2
Headache (Nervous system disorders) | 12
Hydrocephalus (Nervous system disorders) | 1
Intracranial hemorrhage (Nervous system disorders) | 1
Lethargy (Nervous system disorders) | 1
Nervous system disorders - Other (Nervous system disorders) | 1
Paresthesia (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 3
Sinus pain (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 2
Tremor (Nervous system disorders) | 1
Agitation (Psychiatric disorders) | 1
Anxiety (Psychiatric disorders) | 5
Confusion (Psychiatric disorders) | 1
Delirium (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 3
Insomnia (Psychiatric disorders) | 3
Acute kidney injury (Renal and urinary disorders) | 7
Chronic kidney disease (Renal and urinary disorders) | 2
Hematuria (Renal and urinary disorders) | 4
Proteinuria (Renal and urinary disorders) | 7
Urinary frequency (Renal and urinary disorders) | 1
Urinary incontinence (Renal and urinary disorders) | 1
Urinary tract pain (Renal and urinary disorders) | 1
Genital edema (Reproductive system and breast disorders) | 1
Menorrhagia (Reproductive system and breast disorders) | 1
Perineal pain (Reproductive system and breast disorders) | 1
Vaginal hemorrhage (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 7
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 11
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 3
Sore throat (Respiratory, thoracic and mediastinal disorders) | 3
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 3
Dry skin (Skin and subcutaneous tissue disorders) | 2
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Purpura (Skin and subcutaneous tissue disorders) | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 8
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 4
Skin ulceration (Skin and subcutaneous tissue disorders) | 1
Flushing (Vascular disorders) | 1
Hypertension (Vascular disorders) | 5
Hypotension (Vascular disorders) | 9
Peripheral ischemia (Vascular disorders) | 1
Vascular disorders - Other (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Daunorubicin Hydrochloride, Cytarabine, Dasatinib) (N=61)
Anemia (Blood and lymphatic system disorders) | 58
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 5
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 8
Febrile neutropenia (Blood and lymphatic system disorders) | 47
Leukocytosis (Blood and lymphatic system disorders) | 6
Lymph node pain (Blood and lymphatic system disorders) | 3
Atrioventricular block first degree (Cardiac disorders) | 2
Cardiac disorders - Other (Cardiac disorders) | 5
Chest pain - cardiac (Cardiac disorders) | 2
Heart failure (Cardiac disorders) | 3
Left ventricular systolic dysfunction (Cardiac disorders) | 3
Mitral valve disease (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 5
Sinus bradycardia (Cardiac disorders) | 3
Sinus tachycardia (Cardiac disorders) | 16
Ventricular arrhythmia (Cardiac disorders) | 2
Ear and labyrinth disorders - Other (Ear and labyrinth disorders) | 1
Hypothyroidism (Endocrine disorders) | 1
Blurred vision (Eye disorders) | 6
Conjunctivitis (Eye disorders) | 3
Eye disorders - Other (Eye disorders) | 3
Eye pain (Eye disorders) | 2
Floaters (Eye disorders) | 1
Keratitis (Eye disorders) | 2
Photophobia (Eye disorders) | 2
Retinal vascular disorder (Eye disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 12
Anal hemorrhage (Gastrointestinal disorders) | 2
Anal pain (Gastrointestinal disorders) | 2
Ascites (Gastrointestinal disorders) | 2
Bloating (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 30
Dental caries (Gastrointestinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 44
Dyspepsia (Gastrointestinal disorders) | 3
Dysphagia (Gastrointestinal disorders) | 5
Enterocolitis (Gastrointestinal disorders) | 1
Fecal incontinence (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 4
Gastric hemorrhage (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 9
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 8
Gastrointestinal pain (Gastrointestinal disorders) | 1
Gingival pain (Gastrointestinal disorders) | 2
Hemorrhoids (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 24
Nausea (Gastrointestinal disorders) | 47
Oral hemorrhage (Gastrointestinal disorders) | 2
Oral pain (Gastrointestinal disorders) | 8
Rectal hemorrhage (Gastrointestinal disorders) | 1
Rectal pain (Gastrointestinal disorders) | 4
Rectal ulcer (Gastrointestinal disorders) | 1
Stomach pain (Gastrointestinal disorders) | 2
Tooth discoloration (Gastrointestinal disorders) | 1
Toothache (Gastrointestinal disorders) | 3
Typhlitis (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 37
Chills (General disorders) | 12
Edema face (General disorders) | 3
Edema limbs (General disorders) | 19
Edema trunk (General disorders) | 1
Facial pain (General disorders) | 1
Fatigue (General disorders) | 47
Fever (General disorders) | 26
General disorders and administration site conditions - Other (General disorders) | 10
Infusion related reaction (General disorders) | 4
Injection site reaction (General disorders) | 1
Localized edema (General disorders) | 3
Malaise (General disorders) | 3
Non-cardiac chest pain (General disorders) | 7
Pain (General disorders) | 5
Cholecystitis (Hepatobiliary disorders) | 1
Anorectal infection (Infections and infestations) | 1
Catheter related infection (Infections and infestations) | 3
Device related infection (Infections and infestations) | 4
Enterocolitis infectious (Infections and infestations) | 1
Infections and infestations - Other (Infections and infestations) | 14
Lip infection (Infections and infestations) | 2
Lung infection (Infections and infestations) | 12
Lymph gland infection (Infections and infestations) | 1
Mucosal infection (Infections and infestations) | 2
Paronychia (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1
Sepsis (Infections and infestations) | 3
Sinusitis (Infections and infestations) | 3
Skin infection (Infections and infestations) | 6
Soft tissue infection (Infections and infestations) | 1
Tooth infection (Infections and infestations) | 1
Upper respiratory infection (Infections and infestations) | 3
Urinary tract infection (Infections and infestations) | 3
Vaginal infection (Infections and infestations) | 2
Vulval infection (Infections and infestations) | 1
Wound infection (Infections and infestations) | 1
Bruising (Injury, poisoning and procedural complications) | 10
Fall (Injury, poisoning and procedural complications) | 3
Injury, poisoning and procedural complications - Other (Injury, poisoning and procedural complications) | 1
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 1
Activated partial thromboplastin time prolonged (Investigations) | 18
Alanine aminotransferase increased (Investigations) | 41
Alkaline phosphatase increased (Investigations) | 21
Aspartate aminotransferase increased (Investigations) | 30
Blood bilirubin increased (Investigations) | 19
Cardiac troponin I increased (Investigations) | 1
Cholesterol high (Investigations) | 1
Creatinine increased (Investigations) | 10
Ejection fraction decreased (Investigations) | 1
Electrocardiogram QT corrected interval prolonged (Investigations) | 15
Fibrinogen decreased (Investigations) | 2
INR increased (Investigations) | 22
Investigations - Other (Investigations) | 1
Lymphocyte count decreased (Investigations) | 32
Lymphocyte count increased (Investigations) | 8
Neutrophil count decreased (Investigations) | 51
Platelet count decreased (Investigations) | 51
Weight gain (Investigations) | 3
Weight loss (Investigations) | 12
White blood cell decreased (Investigations) | 40
Anorexia (Metabolism and nutrition disorders) | 27
Dehydration (Metabolism and nutrition disorders) | 1
Hypercalcemia (Metabolism and nutrition disorders) | 5
Hyperglycemia (Metabolism and nutrition disorders) | 40
Hyperkalemia (Metabolism and nutrition disorders) | 10
Hypermagnesemia (Metabolism and nutrition disorders) | 7
Hypernatremia (Metabolism and nutrition disorders) | 5
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1
Hyperuricemia (Metabolism and nutrition disorders) | 14
Hypoalbuminemia (Metabolism and nutrition disorders) | 38
Hypocalcemia (Metabolism and nutrition disorders) | 36
Hypoglycemia (Metabolism and nutrition disorders) | 8
Hypokalemia (Metabolism and nutrition disorders) | 30
Hypomagnesemia (Metabolism and nutrition disorders) | 14
Hyponatremia (Metabolism and nutrition disorders) | 30
Hypophosphatemia (Metabolism and nutrition disorders) | 20
Metabolism and nutrition disorders - Other (Metabolism and nutrition disorders) | 4
Tumor lysis syndrome (Metabolism and nutrition disorders) | 1
Abdominal soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 6
Arthritis (Musculoskeletal and connective tissue disorders) | 3
Avascular necrosis (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 15
Bone pain (Musculoskeletal and connective tissue disorders) | 5
Buttock pain (Musculoskeletal and connective tissue disorders) | 3
Chest wall pain (Musculoskeletal and connective tissue disorders) | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 10
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 10
Neck pain (Musculoskeletal and connective tissue disorders) | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Akathisia (Nervous system disorders) | 1
Amnesia (Nervous system disorders) | 2
Ataxia (Nervous system disorders) | 1
Concentration impairment (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 15
Dysgeusia (Nervous system disorders) | 5
Headache (Nervous system disorders) | 31
Lethargy (Nervous system disorders) | 2
Memory impairment (Nervous system disorders) | 1
Nervous system disorders - Other (Nervous system disorders) | 1
Peripheral motor neuropathy (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 4
Tremor (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 13
Confusion (Psychiatric disorders) | 1
Delirium (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 11
Hallucinations (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 15
Acute kidney injury (Renal and urinary disorders) | 1
Chronic kidney disease (Renal and urinary disorders) | 5
Hematuria (Renal and urinary disorders) | 4
Proteinuria (Renal and urinary disorders) | 9
Renal and urinary disorders - Other (Renal and urinary disorders) | 1
Urinary frequency (Renal and urinary disorders) | 2
Breast pain (Reproductive system and breast disorders) | 1
Genital edema (Reproductive system and breast disorders) | 1
Menorrhagia (Reproductive system and breast disorders) | 3
Reproductive system and breast disorders - Other (Reproductive system and breast disorders) | 3
Vaginal discharge (Reproductive system and breast disorders) | 1
Vaginal hemorrhage (Reproductive system and breast disorders) | 2
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 4
Apnea (Respiratory, thoracic and mediastinal disorders) | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 3
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 22
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 26
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 8
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 5
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 9
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 13
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 3
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 5
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 6
Alopecia (Skin and subcutaneous tissue disorders) | 8
Dry skin (Skin and subcutaneous tissue disorders) | 5
Erythema multiforme (Skin and subcutaneous tissue disorders) | 3
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2
Pain of skin (Skin and subcutaneous tissue disorders) | 2
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 4
Periorbital edema (Skin and subcutaneous tissue disorders) | 1
Photosensitivity (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 8
Purpura (Skin and subcutaneous tissue disorders) | 5
Rash acneiform (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 31
Scalp pain (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 18
Skin ulceration (Skin and subcutaneous tissue disorders) | 3
Flushing (Vascular disorders) | 1
Hematoma (Vascular disorders) | 5
Hypertension (Vascular disorders) | 14
Hypotension (Vascular disorders) | 14
Thromboembolic event (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less